CLINICAL TRIAL: NCT00118092
Title: A Phase II Trial of 17-Allylamino-17-Demethoxygeldanamycin (17-AAG) in Patients With Hormone-Refractory Metastatic Prostate Cancer
Brief Title: 17-AAG in Treating Patients With Metastatic Prostate Cancer That Did Not Respond to Previous Hormone Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01466; NCI-2012-01466 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MAYO-MC0453; NCI-6651; CDR0000433492; MC0453 (Other: Mayo Clinic); 6651 (Other: CTEP); N01CM62205 (NIH)
Record Dates: First submitted 2005-07-08; First posted 2005-07-11 (Estimated); Results first posted 2017-02-20 (Actual); Last update posted 2017-04-18 (Actual); Status verified 2017-03

CONDITIONS: Adenocarcinoma of the Prostate; Recurrent Prostate Cancer; Stage IV Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — tanespimycin

ARMS (1):
- Treatment (tanespimycin) (Experimental): Patients receive 17-N-allylamino 17-demethoxygeldanamycin (17-AAG) IV over 2-6 hours on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients who achieve a complete response (CR) receive 2 additional courses of treatment beyond documentation of CR.
  Interventions: Drug: tanespimycin; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: tanespimycin — Given IV
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well 17-AAG works in treating patients with metastatic prostate cancer that did not respond to previous hormone therapy. Drugs used in chemotherapy, such as 17-AAG, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the prostate-specific antigen (PSA) response in patients with hormone-refractory metastatic prostate cancer treated with 17-N-allylamino-17-demethoxygeldanamycin (17-AAG).

SECONDARY OBJECTIVES:

I. Determine the overall survival and disease-free survival rate in patients treated with this drug.

II. Determine the safety profile of this drug in these patients. III. Determine the duration of PSA response and PSA control in patients treated with this drug.

IV. Determine the partial and complete response rates in patients with measurable disease treated with this drug.

V. Correlate changes in expression levels of interleukin-6, maspin, and NF-kappaB in serum and tissue with cancer and treatment-related outcomes in patients treated with this drug.

OUTLINE: This is a multicenter study. Patients receive 17-N-allylamino-17-demethoxygeldanamycin (17-AAG) IV over 2-6 hours on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients who achieve a complete response (CR) receive 2 additional courses of treatment beyond documentation of CR.

After completion of study treatment, patients are followed every 3 months for 1 year and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 16-28 patients will be accrued for this study within 20 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate

  * Metastatic disease
* Measurable or evaluable disease

  * Prostate-specific antigen (PSA) ≥ 5 ng/mL OR new areas of bony metastases on bone scan are required for patients with no measurable disease
* Objective disease progression OR rising PSA despite receiving androgen deprivation therapy and undergoing antiandrogen withdrawal

  * Patients with a rising PSA must have 2 successive elevations (measured ≥ 1 week apart)
* Must be castrate (testosterone < 50 ng/mL)

  * Luteinizing hormone-releasing hormone agonist therapy must be continued during study participation to maintain castrate levels of testosterone
* Must have received ≥ 1 prior chemotherapy regimen for metastatic disease
* No known brain metastases requiring active therapy

  * Previously treated asymptomatic brain metastases allowed
* Performance status - ECOG 0-2
* At least 12 weeks
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 8.0 g/dL
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* SGOT and/or SGPT ≤ 2.5 times ULN AND alkaline phosphatase normal
* Alkaline phosphatase ≤ 4 times ULN AND SGOT and/or SGPT normal
* Creatinine clearance ≥ 60 mL/min
* Creatinine normal
* QTc < 450 msec for male patients
* LVEF > 40% by MUGA
* EF normal by MUGA if prior anthracycline therapy
* No congenital long QT syndrome
* No left bundle branch block
* Deep venous thrombosis or other clinically significant thromboembolic event within the past 6 months allowed provided patient is clinically stable on anticoagulation therapy
* No history of serious ventricular arrhythmia (i.e., ventricular tachycardia or ventricular fibrillation ≥ 3 beats in a row)
* No myocardial infarction within the past year
* No cerebrovascular accident or transient ischemic attack within the past 6 months
* No New York Heart Association class III or IV congestive heart failure
* No poorly controlled angina
* No uncontrolled dysrhythmia or dysrhythmias requiring medication
* No active ischemic heart disease within the past 12 months
* No other significant cardiac disease
* Pulmonary embolus allowed within the past 6 months provided patient is clinically stable on anticoagulation therapy
* Fertile patients must use effective contraception
* Willing and able to provide blood samples
* No serious allergy (i.e., hypotension, dyspnea, anaphylaxis, or edema) to eggs
* No other concurrent malignancy or history of a curatively treated malignancy with a survival prognosis of < 5 years
* No known HIV positivity
* No active infection
* No other severe acute or chronic medical or psychiatric condition or laboratory abnormality that would preclude study participation
* At least 4 weeks since prior flutamide (6 weeks for bicalutamide or nilutamide)
* At least 28 days since prior radiotherapy
* No prior radiotherapy field that included the heart (e.g., mantle)
* More than 6 months since prior coronary or peripheral artery bypass grafting
* More than 28 days since prior investigational agents for prostate cancer
* No concurrent agents that interact with cytochrome P450 3A4
* No concurrent warfarin for anticoagulation

  * Concurrent low molecular weight heparin injection allowed
* No concurrent medications that would prolong QTc
* No other concurrent antineoplastic agents
* Concurrent zoledronate for bone metastases or hypercalcemia allowed

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2005-01; Primary Completion 2006-05 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Heath, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Tanespimycin): Patients receive 300 mg/m^2 17-N-allylamino 17-demethoxygeldanamycin (17-AAG) IV over 2-6 hours on days 1, 8, and 15. > Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Treatment (Tanespimycin)
Started | 17
Completed | 15
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Tanespimycin)
Number analyzed (Participants) | 15
Age, Continuous [Median (Full Range); unit: years] | 68 [52 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: PSA Response as Defined by the Recommendations of the Prostate-Specific Antigen Working Group
Description: Normalization: PSA ≤4.0 ng/ml. This must be confirmed by a second PSA value measured when patient returns in 4-6 weeks. This qualifies as a CR response. > > 50% decline: A 50% decline in PSA value from baseline which must be confirmed by a second PSA value measured when patient returns in 4-6 weeks later. This qualifies as a PR response.>
  > Progression: A 25% or greater increase over baseline and an increase in the PSA level by at least 5 ng/mL, which is confirmed by a second value obtained approximately one week later. In addition, radiographic scans are required to confirm that a disease progression is by PSA only.
Time Frame: Up to 1 year
Population: All 15 eligible patients that started treatment were evaluated.
Measure: Number; unit: participants
Arm/Group | Treatment (Tanespimycin)
Number analyzed (Participants) | 15
participants | 0

2. Secondary Outcome: Proportion of Overall Responses
Description: Confirmed response rate was defined using Response Evaluation Criteria In Solid Tumors (RECIST). A confirmed response is defined as a complete response (CR) or partial response (PR) observed on subsequent scans at least 4 weeks apart. Confirmed response rate was estimated by the number of successes divided by the total number of evaluable patients. Complete Response (CR) is defined as the disappearance of all target lesions. Partial Response (PR) is defined as a 30% decrease in sum of longest diameter of target lesions.
  The proportion of confirmed responses will be estimated by the number of patients with confirmed responses divided by the total number of evaluable patients. Ninety-five percent confidence intervals for the true success proportion will be calculated according to the approach of Duffy and Santner.
Time Frame: Up to 3 years
Population: All 15 eligible patients that started treatment were evaluated.
Measure: Number (95% Confidence Interval); unit: percentage of responses
Arm/Group | Treatment (Tanespimycin)
Number analyzed (Participants) | 15
percentage of responses | 0 [0 to 22]

3. Secondary Outcome: Overall Survival
Description: Overall survival time is defined as the time from registration to death due to any cause. The distribution of survival time will be estimated using the method of Kaplan-Meier.
Time Frame: From registration to death due to any cause, assessed up to 3 years
Population: All 15 eligible patients that started treatment were evaluated.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Tanespimycin)
Number analyzed (Participants) | 15
months | 9.4 [2.7 to 17.7]

4. Secondary Outcome: Disease-free Survival
Description: Disease-free survival time is defined as the time from registration to documentation of disease progression. If a patient dies without a documentation of disease progression, the patient will be considered to have had progressed at the time of their death. In patients who have achieved a PSA response, we will assess the time to PSA progression. If the patient is declared to be a major treatment violation, the patient will be censored on the date the treatment violation was declared to have occurred. In the case of a patient starting treatment and then never returning for any evaluations, the patient will be censored for progression on day 1 post-registration. The distribution of disease-free survival time will be estimated using the method of Kaplan-Meier.
Time Frame: From registration to documentation of disease progression, assessed up to 3 years
Population: All 15 eligible patients that started treatment were evaluated.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Tanespimycin)
Number analyzed (Participants) | 15
months | 1.8 [1.3 to 3.4]

5. Secondary Outcome: Duration of PSA Response and PSA Control
Description: The distribution of this response duration will be estimated using the method of Kaplan-Meier. In patients whose PSA has declined from baseline by at least 30 %, "duration of PSA response" will be defined as the time from PSA response to time of progression. If a patient goes on to alternate therapy, they will be censored at the date they end treatment on this study. "Duration of PSA Control" is defined as the time from the date of the first 30% decline in PSA until an inflection point is identified. Inflection point is defined as the time to first consistent PSA increase, the point at which PSA began what becomes a continuous increase
  > (retrospectively identified). The inflection point is the point at which disease control could assume to be lost.
Time Frame: From PSA response to time of progression, assessed up to 1 year
Population: No participants with PSA response or PSA control.
Arm/Group | Treatment (Tanespimycin)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Groups:
- Treatment (Tanespimycin): Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | Treatment (Tanespimycin)
Serious Adverse Events (participants affected / at risk) | 2/17
Other Adverse Events (participants affected / at risk) | 16/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Tanespimycin) (N=17)
Neutrophil count decreased (Investigations) | 1 (2)
Thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Tanespimycin) (N=17)
Hemoglobin decreased (Blood and lymphatic system disorders) | 14 (19)
Premature ventricular contractions (Cardiac disorders) | 1 (2)
Sinus arrhythmia (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Supraventricular extrasystoles (Cardiac disorders) | 3 (4)
Vision blurred (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (4)
Constipation (Gastrointestinal disorders) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 6 (6)
Flatulence (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 8 (10)
Vomiting (Gastrointestinal disorders) | 4 (6)
Fatigue (General disorders) | 10 (15)
Fever (General disorders) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 4 (6)
Alkaline phosphatase increased (Investigations) | 7 (10)
Aspartate aminotransferase increased (Investigations) | 8 (10)
Electrocardiogram QTc interval prolonged (Investigations) | 2 (2)
Leukocyte count decreased (Investigations) | 2 (3)
Lymphocyte count decreased (Investigations) | 5 (5)
Neutrophil count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 4 (6)
Weight loss (Investigations) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 6 (7)
Blood glucose increased (Metabolism and nutrition disorders) | 7 (13)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Serum albumin decreased (Metabolism and nutrition disorders) | 8 (11)
Serum calcium decreased (Metabolism and nutrition disorders) | 3 (5)
Serum phosphate decreased (Metabolism and nutrition disorders) | 1 (2)
Serum potassium decreased (Metabolism and nutrition disorders) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Headache (Nervous system disorders) | 2 (3)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Hemorrhage urinary tract (Renal and urinary disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Body odor (Skin and subcutaneous tissue disorders) | 3 (4)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less